CLINICAL TRIAL: NCT02863523
Title: COMRADE: Collaborative Care Management for Distress and Depression in Rural Diabetes
Acronym: COMRADE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Doyle M. Cummings, Professor of Family Medicine, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COMRADE
Record Dates: First submitted 2016-08-03; First posted 2016-08-11 (Estimated); Results first posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-03

CONDITIONS: Type 2 Diabetes Mellitus; Diabetes-related Distress; Depression
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Integrated Behavioral Intervention (Experimental): Patients receive intensive behavioral counseling that may include elements of cognitive behavioral therapy, problem solving therapy, and small changes lifestyle counseling in addition to medical care.
  Interventions: Behavioral: Integrated Behavioral Care
- Usual Care (No Intervention): Patients receive usual care

INTERVENTIONS:
Behavioral: Integrated Behavioral Care — Patients receive intensive behavioral counseling that may include elements of cognitive behavioral therapy, problem solving therapy, and small changes lifestyle counseling in addition to medical care.
  Arms: Integrated Behavioral Intervention

SUMMARY:
The study will implement and evaluate, using a pragmatic comparative effectiveness trial, a unique collaborative, stepped-care intervention for patients with uncontrolled Type 2 diabetes and co-morbid distress and/or depression.

DETAILED DESCRIPTION:
The investigators plan to implement and evaluate, using a pragmatic comparative effectiveness trial, a unique collaborative, stepped-care intervention for patients with uncontrolled Type 2 diabetes and co-morbid distress and/or depression. The investigators approach will combine practice-based medical and cognitive behavioral treatment with strong community-based support to immediately place the patient at the right level of intervention based on disease and severity and to step-up treatment intensity and follow-up if the initial response is inadequate. The practice-based component will use a care manager linked to medical, pharmacologic, and behavioral colleagues. The community based component will utilize community health workers to provide support and facilitate access to resources. Goals include: 1) implementing and evaluating the effectiveness of this intervention; 2) examining the impact of this approach on psychological mediators of improved glycosylated hemoglobin (HbA1c); and 3) building, sustaining, and disseminating a cost-effective care model.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical Diagnosis of Type 2 diabetes mellitus
2. Glycosylated Hemoglobin (HbA1c) > 7.0 = Uncontrolled
3. Positive score on diabetes related distress 2 question screener and/or
4. Positive score on Patient Health Questionnaire (PHQ-2) 2 question screener

Exclusion Criteria: a diagnosis [from billing records using International Classification of Disease, 9th Edition (ICD-9) codes] of:

1. advanced disease (e.g., end stage renal disease, advanced heart failure, blindness, metastatic cancer and including those who are in active treatment for cancer), or
2. alcoholism or
3. cognitive impairment, or
4. major psychiatric disease or
5. any type of physical or mental impairment that would preclude active participation

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2014-09; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- East Carolina University, Greenville, North Carolina, United States

REFERENCES:
- [Background] Cummings DM, Lutes LD, Littlewood K, Solar C, Carraway M, Kirian K, Patil S, Adams A, Ciszewski S, Edwards S, Gatlin P, Hambidge B. Randomized Trial of a Tailored Cognitive Behavioral Intervention in Type 2 Diabetes With Comorbid Depressive and/or Regimen-Related Distress Symptoms: 12-Month Outcomes From COMRADE. Diabetes Care. 2019 May;42(5):841-848. doi: 10.2337/dc18-1841. Epub 2019 Mar 4. PMID 30833367
- [Background] Lutes LD, Cummings DM, Littlewood K, Le MT, Kirian K, Patil S, Solar C, Carraway M, Hambidge B. A Tailored Cognitive-Behavioural Intervention Produces Comparable Reductions in Regimen-Related Distress in Adults With Type 2 Diabetes Regardless of Insulin Use: 12-Month Outcomes From the COMRADE Trial. Can J Diabetes. 2020 Aug;44(6):530-536. doi: 10.1016/j.jcjd.2020.05.016. Epub 2020 Jun 10. PMID 32792107
- [Result] Lutes LD, Cummings DM, Littlewood K, Solar C, Carraway M, Kirian K, Patil S, Adams A, Ciszewski S, Hambidge B. COMRADE: A randomized trial of an individually tailored integrated care intervention for uncontrolled type 2 diabetes with depression and/or distress in the rural southeastern US. Contemp Clin Trials. 2018 Jul;70:8-14. doi: 10.1016/j.cct.2018.04.007. Epub 2018 Apr 20. PMID 29680319

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Integrated Behavioral Intervention | Usual Care
Started | 67 | 72
Completed | 67 | 72
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Integrated Behavioral Intervention | Usual Care | Total
Number analyzed (Participants) | 67 | 72 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.67 (9.67) | 54.71 (9.3) | 53.7 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 55 | 108
  Male | 14 | 17 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 53 | 48 | 101
  White or mixed race | 14 | 24 | 38
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 67 | 72 | 139
HbA1c [Mean (Standard Deviation); unit: percent] | 9.8 (2.1) | 9.3 (1.7) | 9.6 (1.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (%)
Description: Change from baseline in HbA1c or glycosylated hemoglobin (%)
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: change from baseline in A1c (%)
Arm/Group | Integrated Behavioral Intervention | Usual Care
Number analyzed (Participants) | 67 | 72
change from baseline in A1c (%) | -0.92 (1.8) | -0.31 (2.0)

2. Secondary Outcome: Change From Baseline in Diabetes Regimen-Related Distress
Description: Diabetes regimen-related distress is a measure of the emotional response to having and managing diabetes and is measured by a subscale of 5 items (#5, 6, 10, 12, 16) from the Diabetes-related Distress instrument (DDS-17). Each item is rated from 1 (not a problem) - 6 (very serious problem) and therefore the total score for this sub-score ranges from 5 - 30. The mean score for an individual can be computed as the sum of the 5 items divided by 5. For this study outcome, the investigators computed the average change (increase or decrease) in the mean RRD score from baseline to 12-mo. follow-up.
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrated Behavioral Intervention | Usual Care
Number analyzed (Participants) | 67 | 72
score on a scale | -1.1 (1.0) | -0.3 (1.2)
Statistical Analysis 1: Comparison: Integrated Behavioral Intervention vs Usual Care; Test type: Superiority; p < 0.0001, t-test, 2 sided

3. Other Pre Specified Outcome: Change in Diabetes Self-care Activities
Description: Diabetes self-care activities as measured by the Self-reported Diabetes Self Care Activities (SDSCA) instrument. The SDSCA is a questionnaire which assesses levels of self-care in adults with diabetes. The tool contains 11 items, which measure the frequency of performing diabetes self-care activities over the last seven days including diet, exercise, blood glucose testing, foot care and tobacco use. The respondent marks the number of days on which the indicated behavior was performed on an eight-point Likert scale (0 - 7) to answer the questions. The first ten items are summed to a total score. The eleventh item focuses on smoking habits and assesses the average number of cigarettes smoked per day. For the present study, the total score was summed and divided by 11 items to create a mean score and then the average change from baseline to 12 month follow-up.
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrated Behavioral Intervention | Usual Care
Number analyzed (Participants) | 67 | 72
score on a scale | 1.1 (1.3) | 0.58 (1.4)
Statistical Analysis 1: Comparison: Integrated Behavioral Intervention vs Usual Care; Test type: Superiority; p < 0.03, t-test, 2 sided

4. Other Pre Specified Outcome: Change in Depressive Symptoms
Description: Change in depressive symptoms as measured by the Patient Health Questionnaire-9 (PHQ-9) instrument for depressive symptoms. Diagnosis based on Total PHQ-9 Score; Interpretation:
  Minimal depression 0-4 Mild depression 5-9 Moderate depression 10-14 Moderately severe depression 15-19 Severe depression 20-27
Time Frame: Baseline to 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integrated Behavioral Intervention | Usual Care
Number analyzed (Participants) | 67 | 72
score on a scale | -3.4 (5.0) | -0.9 (6.2)
Statistical Analysis 1: Comparison: Integrated Behavioral Intervention vs Usual Care; Test type: Superiority; p < 0.01, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Integrated Behavioral Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/72
Other Adverse Events (participants affected / at risk) | 0/67 | 0/72

LIMITATIONS AND CAVEATS:
Adverse event detection was limited to events potentially associated with behavioral counseling.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-11): https://cdn.clinicaltrials.gov/large-docs/23/NCT02863523/Prot_SAP_000.pdf